CLINICAL TRIAL: NCT06817252
Title: Effects of a Mediterranean Dietary Pattern With White Potato on Cardiometabolic Health in Adults With Pre-Diabetes
Brief Title: How a Mediterranean Diet With Potatoes Impacts Heart and Metabolic Health in Adults With Pre-Diabetes
Acronym: MEDPOT-PREDM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNLV-2024-385
Record Dates: First submitted 2025-01-24; First posted 2025-02-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-01

CONDITIONS: Prediabetes; Lipid Profile; Hypertension; Glycemic Control; Arterial Stiffness, Blood Pressure; Inflammation Biomarkers; Dietary Quality; Body Composition Measurement; Waist Circumference; Anthropometrics: Height and Weight
Keywords: White Potato; Prediabetes; Mediterranean Diet; Cardiometabolic Health; Dietary Quality
MeSH Terms: conditions — Prediabetic State; Hypertension; Body Weight

STUDY DESIGN:
Intervention Model Description: This study does not involve aType of Drug, Biological/Vaccine, or Combination Product. This is a behavioral intervention focusing on a Mediterranean Diet Nutrition Education with or without baked potatoes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet Nutrition Education (Active Comparator)
  Interventions: Behavioral: Mediterranean Diet Nutrition Education
- Mediterranean Diet Nutrition Education with Baked White Potatoes (Experimental)
  Interventions: Behavioral: Mediterranean Diet Nutrition Education with Baked White Potato

INTERVENTIONS:
Behavioral: Mediterranean Diet Nutrition Education — Participants randomized to receive the Mediterranean Diet Nutrition Education will receive a pre-recorded education session (lasting approximately 1 hour) they can watch at home after their Baseline and 6-Week Study Visits, which will be created by the PI and Co-I's of the study (who are comprised of Professors who are either Registered Dietitian credentialed or have experience with creating nutrition/physical activity programs), including an explanation of the principles and components of a Mediterranean dietary pattern and its benefits, guidance on recommended intake of various food groups, budget-friendly strategies for incorporation, supporting resources (educational materials and online tools), and techniques for overcoming barriers to following a Mediterranean dietary pattern. Additional educational materials will be provided to participants through computer or web-based sources.
  Arms: Mediterranean Diet Nutrition Education
Behavioral: Mediterranean Diet Nutrition Education with Baked White Potato — Participants randomized to receive the Mediterranean Diet Nutrition Education with Baked White Potatoes will similarly receive a pre-recorded education session (lasting approximately 1 hour) they can watch at home after their Baseline and 6-Week Study Visits (same as the Mediterranean Diet Nutrition Education group). They will also receive will 100 g roasted white russet potatoes with the skin and will be asked to consume the regimen as a part of their meals (breakfast, lunch, dinner) or as a snack throughout the day to contribute to a balanced meal plan. The baked white potato regimen will be pre-portioned (in 100g amounts), stored in the freezer and given in freezer-microwave safe containers. The baked white potato regimen is approximately 100 kilocalories, 22g carbohydrates, and 0.2g of fat . In order to increase participants' compliance, they will be informed of a variety of ways to consume the baked white potato regimen.
  Arms: Mediterranean Diet Nutrition Education with Baked White Potatoes

SUMMARY:
The goal of this clinical trial is to is to determine the effects of baked potato with the skin (BP) + nutrition education focused on adherence for a Mediterranean Dietary Pattern (MEDNE) on glycemic control, cardiometabolic health, and dietary quality in individuals with pre-diabetes from different demographic backgrounds. The main questions it aims to answer are:

* Does BP+MEDNE contribute to improvements in indices of glycemic control, vascular function, blood lipids, inflammation/oxidative stress, and body composition?
* Does BP+MEDNE contribute to improvements to overall dietary intake and quality?

Researchers will compare BP+MEDNE to MEDNE alone to see if BP+MEDNE can improve glycemic control, cardiometabolic health, and dietary quality in individuals with pre-diabetes from different demographic backgrounds.

Participants will:

* Be asked to come to the study site initially for a Screening Study Visit to confirm eligibility.
* Be asked to come the study site for a Pre-Baseline and Pre-12-Week Study Visit (one week prior to Baseline and 12-Week Study Visits) for placement of placement of a continuous glucose monitor and wearable devices to be removed at Baseline and 12-Week Study Visits.
* Be asked to come to the study site for Baseline, 6- and 12-Week Study Visits for assessments of glycemic control and cardiometabolic health.
* Be asked to complete 3-Day Food Records throughout the 12 week study period for assessment of dietary quality (5 total)
* Receive pre-recorded MEDNE ( which can be accessed via computer device/ipad/smartphone) after Baseline and 6-Week Study Visits.
* If randomized to the BP+MEDNE group, participants will receive pre-prepared baked potatoes with the skin for the 12-week study period (every 3 weeks) at Baseline and 6-Week Study Visits and asked to come to the study site for picking up the pre-prepared baked potatoes at weeks 3 and 9 of the study period.

DETAILED DESCRIPTION:
Study Overview: Investigators will recruit 60 adults with pre-diabetes from different demographic backgrounds, between the ages of 45 and 80 years to participate in a 12-week randomized controlled trial (RCT) examining baked potato with the skin (BP) + nutrition education focused on adherence for a Mediterranean Dietary Pattern (MEDNE) compared to MEDNE alone. Potential participants will be recruited from the metropolitan Las Vegas area through campus and community advertisements including flyers, newspaper articles, social media, and public events. Investigators will randomize eligible, consenting participants to receive either the BP+MEDNE or MEDNE in a 1:1 ratio. Investigators will use a computer-generated randomization method to manage the random assignment of either group.

Prescreen Interview: Potential participants who inquire about the study by calling the recruitment phone line, will be given a brief overview of the study and will be pre-screened by telephone interview to determine whether they should be invited for the in-person screening visit. Eligibility will be based on inclusion/exclusion criteria and responses to questions about medical history and dietary habits. Potential participants will be invited to report to the clinical facilities in the Health Sciences Building at UNLV (study site) for their first on-site visit (and all subsequent visits if the participant qualifies) to ascertain eligibility (screening study visit). This pre-screening interview will occur prior to participants consenting (which occurs at the in person screening study visit).

Screening Study Visit: Potential participants who inquire about the study by calling the recruitment phone line will be given a brief overview of the study and pre-screened by telephone to determine whether they should be invited for the in-person screening visit. Eligibility will be based on inclusion/exclusion criteria and responses to questions about medical and diet history during the pre-screen phone interview. Potentially eligible participants will be invited to report to the study site for their first on-site visit for screening (and all subsequent visits if the participant qualifies) to ascertain eligibility (Screening Study Visit). During the first in-person study visit for screening, the potential participants will be provided with verbal and written explanations of the project and will have any questions regarding the study answered by trained research personnel during the informed consent process. Consenting participants will be asked to sign an informed consent document (with a copy provided to the participant to take home). To confirm eligibility, the Screening Study Visit will consist of measurements of HbA1c (Afinion HbA1c Point of Care) via finger stick blood draw to confirm pre-diabetes, in addition to anthropometrics, blood pressure, and questions regarding medical history and medication use (fasting blood glucose via ACCU-CHECK Glucometer will be assessed but not as an eligibility criteria). Potential participants will also complete a 7-day food frequency questionnaire, to indicate whether individuals frequently consume baked white potatoes. If participants are considered "non-frequent" white potato consumers, they will be included in the study and asked to come for subsequent visits and study visits. Participants who are not eligible will be thanked for their time and participation and told the specific reasoning for why they do not meet the inclusion criteria. Eligible participants will be asked to complete a three-day food record using NCI's Automated Self-Administered 24-Hour Dietary Assessment Tool to assess typical dietary intake and dietary quality (Healthy Eating Index [HEI]-2020 scoring), prior to their Baseline Study Visit at participants homes via a computer, ipad, or smartphone. The Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24) is a web-based dietary recall system developed by the National Cancer Institute. It allows participants to self-report their dietary intake over the past 24 hours using a user-friendly interface that prompts for detailed food and beverage consumption. The tool can be distributed via a unique web link provided to participants, enabling remote data collection without requiring in-person visits.

Pre Baseline and 12-Week Visits: One week prior to the Baseline and 12-Week Study Visits, eligible participants will be asked to come to the study site to have placement of a continuous glucose monitor from training research staff (Dexcom G7) and wearable devices (ActiGraph Accelerometry) for assessments of real-time blood glucose levels, physical activity, and sleeping patterns. At their Baseline and 12-Week Study Visits, trained research staff will remove the Dexcom CGM from the participant and discard it. Similarly at their Baseline and 12-Week Study Visits, the Actigraph wearable device will be removed from trained research staff.

Baseline, 6- and 12-Week Study Visits: At the Baseline, 6-, and 12-Week Study Visits participants will be asked to come fasted to the study site (between 7:00-10:00 A.M., 12 hours after the abstinence from caffeine and 24 hours after the last bout of moderate/heavy physical activity); vascular assessments (blood pressure, Pulse Wave Velocity, Pulse Wave Analysis) will be measured followed by body composition (Bioelectrical Impedance Analysis), finger prick blood draw (fasting blood glucose and HbA1c), venous blood draw (lipid profiles, inflammatory, and oxidative stress biomarkers), anthropometrics (height, weight, and waist/hip circumference), assessment of fruit and vegetable intake via Raman Spectroscopy, assessment of physical activity patterns (Five-City Project Physical Activity Recall), nutrition knowledge (General Nutrition Knowledge Questionnaire), MD adherence (Mediterranean Diet Adherence Screener), barriers to Mediterranean Diet Adherence (Barrier Analysis Questionnaire), and sleep quality (Pittsburg Sleep Quality Index). After assessments of outcome measurements at Baseline and 6-Week Study Visits (not at the 12-Week Study Visit), participants will be provided with BP+MEDNE or MEDNE (comparative control). All participants will be provided with MEDNE. In addition to all assessments mentioned for all study visits, at the 12-Week Study Visit there will be assessment of dietary and/or nutrition education acceptability and feasibility.

Dietary Assessments Throughout The Study Period (at week 1, 4, 8, and 12): Participants will be asked to complete a three-day food record using NCI's Automated Self-Administered 24-Hour (ASA24) Dietary Assessment Tool to assess typical dietary intake and diet quality (using HEI-202075) during week 1, 4, 8, and 12 of the study period. This food record can be completed at participants' homes via a computer, ipad or smartphone.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women within the Las Vegas/Henderson NV area
* Ages 45-80 years
* BMI between 25-40 kg/m2
* HbA1c between 5.7-6.4%
* Individuals from different demographic backgrounds (i.e., American Indian or Alaska Native, Caucasians, Asian, Black or African-American, Native Hawaiian, Hispanic, Latino or Pacific Islander)
* Individuals who are considered "non-frequent" white potato consumers (<2 servings of baked potatoes/week)
* Individuals from all races, genders, sexual identities, and religions will be included
* Individuals must follow certain guidelines, including avoiding new medications during the study or significant changes to lifestyle factors (e.g. beginning to smoke or exercise more or less than usual)

Exclusion Criteria:

* Individuals with uncontrolled hypertension (≥160/100mmHg), active cancer, asthma, thyroid, kidney, liver, or pancreatic diseases
* Individuals who are currently using insulin, on dialysis, changing/adding hypoglycemic, anti-hypertensive, and hypocholesterolemic medication within ≤3 months (or throughout the study)
* Individuals participating in weight loss programs or another clinical trial
* Individuals who start smoking
* Individuals who have unstable metabolic or chronic diseases
* Individuals who may have allergies to potatoes
* Woman who are currently pregnant, think they may be pregnant, or who is nursing cannot participate (women must be postmenopausal)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HemoglobinA1c | Baseline and 12-Week Study Visits: 12 weeks
  Fasting HemoglobinA1C percentage measured via Afinion AS100 Analyzer (point of care device)
Change in Blood Glucose Levels | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Fasting Blood Glucose Levels Measured with a Glucometer
Change in Plasma Insulin Levels | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Fasting Plasma Insulin Levels measured via ELISA

SECONDARY OUTCOMES:
Change in blood pressure | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Fasted diastolic and systolic blood pressure, measured via OMRON automated blood pressure device
Changes in Arterial Stiffness-Pulse Wave Velocity | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Fasted measured of arterial stiffness via carotid-femoral and aortic pulse wave velocity (cfPWV) in meters per second (m/s) (SphygmoCor XCEL).
Changes in Arterial Stiffness-Augmentation Index | Baseline, 6-Week, and 12-Week Study Visits: 12 Weeks
  Fasted measured of arterial stiffness via pulse wave analysis (SphygmoCor XCEL) with measure of Augmentation Index (AIx) expressed as a percentage (%)
Changes in Lipid Profiles | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Measure of fasted lipid profiles (total cholesterol, triglycerides, high-density lipoprotein-cholesterol, low-density lipoprotein-cholesterol) all measured in milligrams per deciliter (mg/dL) via Piccolo Xpress chemistry analyzer
Change in Oxidized-LDL | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Fasted oxidized LDL will be measured via ELISA
Changes in waist and hip circumferences | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Waist and hip circumference changes measured in centimeters.
Change in body fat % | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Body fat % measured via Bioelectrical Impedance Analysis (Seca BIA Platform mBCA 554 Medical Body Composition Analyzer)
Changes in Dietary Quality | Pre-Baseline, and weeks 1, 4, 8, and 12 of the study period: 13 weeks (due to assessment prior to Baseline)
  Dietary Quality measured via Health Eating Index-2020 from three-day food records using NCI's Automated Self-Administered 24-Hour Dietary Assessment Tool. The index score will be from 0-100, with 0 indicating poorest diet quality and 100 excellent.
Changes in Nutrition Knowledge | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Measurements of nutrition knowledge via General Nutrition Knowledge Questionnaire which are general questions used to assess a person's understanding of basic nutrition principles and dietary guidelines.
Changes in Fruit and Vegetable Intake Adherence | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Assessment of fruit and vegetable intake will be measured via Raman Spectroscopy (VeggieMeter)
Changes in Physical Activity Patterns | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Assessment of physical activity patterns via Five-City Project Physical Activity Recall
Changes in Sleep Quality | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Assessment of sleep quality measured via Pittsburg Sleep Quality Index wich is a questionnaire used to assess the quality and patterns of sleep over a one-month period, measuring factors like sleep duration, sleep disturbances, and daytime dysfunction. The scores are typically presented as a global score, ranging from 0 to 21, where higher scores indicate poorer sleep quality.
Changes in Arterial Stiffness- Central Systolic Blood Pressure | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Fasted measured of Central Systolic Blood Pressure (cSBP) measured in mmHg (millimeters of mercury) via SphygmoCor XCEL.
Changes in Arterial Stiffness-Central Pulse Pressure | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Fasted measured of Central Pulse Pressure measured in mmHg (millimeters of mercury) via SphygmoCor XCEL.
Changes in Arterial Stiffness-Augmented Pressure | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Fasted measured of Augmented Pressure measured in mmHg (millimeters of mercury) via SphygmoCor XCEL
Changes in Arterial Stiffness-Subendocardial Viability Ratio | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Fasted measured of arterial stiffness via pulse wave analysis (SphygmoCor XCEL) with measure of Subendocardial Viability Ratio expressed as a percentage (%)
Changes In Arterial Stiffness-Transit Time | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Fasted measured of arterial stiffness via transit in milliseconds (SphygmoCor XCEL).
Changes in body weight | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Body weight will be measured in kilograms with a weighing scale
Changes in Body Mass Index | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Body Mass Index will be assessed with a participants height in meters and body weight in kilograms, in the unit of kg/m2
Assessment of Height | Screening
  Height will be assessed in meters (for assessment of BMI at future visits and inclusion criteria)
Changes in high sensitivity C-Reactive Protein | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Fasted measure of plasma high sensitivity C-Reactive Protein in mg/L measured via ELISA
Changes in tumor necrosis factor-alpha | Baseline, 6-Week, and 12-Week Study Visits: 12 Weeks
  Fasted measure of plasma tumor necrosis factor-alpha in pg/mL measured via ELISA
Changes in soluble intercellular adhesion molecule-1 | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Fasted measure of soluble intercellular adhesion molecule-1 in ng/mL measured via ELISA
Changes In Dietary Intake | Pre-Baseline, and weeks 1, 4, 8, and 12 of the study period: 13 weeks (due to assessment prior to Baseline)
  Dietary intake measured from three-day food records using NCI's Automated Self-Administered 24-Hour Dietary Assessment Tool, will be measured throughout the study period to indicate any changes in overall macro and micro nutrient intake between the treatment and comparative control group.
Changes in Mediterranean Diet Adherence | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Measurements of Mediterranean Diet Adherence (Mediterranean Diet Adherence Screener) which are a set of questions used to evaluate how closely an individual's eating habits align with the principles of the Mediterranean diet.
Changes in barriers to Mediterranean Diet Adherence | Baseline, 6- and 12-Week Study Visits: 12 weeks
  Measurements of barriers to Mediterranean Diet Adherence (Barrier Analysis Questionnaire) which are questions that identifies factors that prevent individuals from fully adhering to the Mediterranean diet, such as cultural, economic, or personal obstacles

OTHER OUTCOMES:
Changes in Glucose Time-in-Range and Peak Glucose | Pre-Baseline and Pre-12-Week Study Visits: 14 days, 7 prior to the Baseline and 12-Week Study Visits
  Glucose Time-in-Range and Peak Glucose (mean, nighttime, and daytime glucose levels, in addition to glucose variability) measured via Continuous Glucose Monitoring (Dexcom G7) which will be assessed in units of milligrams per deciliter (mg/dL) for blood glucose levels throughout the days.
Changes in Physical Activity and Sleeping Patterns via Wearable Device | Pre-Baseline and Pre-12-Week Study Visits: 14 days, 7 prior to the Baseline and 12-Week Study Visits
  Physical Activity and Sleeping Patterns assessed vis wearable device (ActiGraph Accelerometry) which is used to objectively assess physical activity and sleep patterns by measuring movement through sensors that track acceleration. The data collected includes metrics like step count, intensity of activity, and sleep duration or quality.

CONTACTS AND LOCATIONS:
Overall Officials: Neda S Akhavan, PhD, RD, Principal Investigator — University of Nevada, Las Vegas
Locations (2):
- United States (2):
  - Department of Kinesiology and Nutrition Sciences, Las Vegas, Nevada
  - University of Nevada Las Vegas, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared because the study did not obtain participant consent for data sharing, and there are concerns regarding the protection of participant privacy and confidentiality. Additionally, institutional and regulatory policies restrict data sharing, and the data are not intended for broader dissemination.